CLINICAL TRIAL: NCT01231724
Title: A Randomized, Double-Blind, Placebo-Controlled, Cross-Over Trial of Topical Allstate in the Prevention of the Signs and Symptoms of the Acute Response to Nasal Allergen Challenge (CETALY0001)
Brief Title: Topical Allstate and Nasal Allergen Challenge
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: study halted prematurely, prior to enrollment of first participant
Sponsor: University of Chicago (Other)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Responsible Party: Principal Investigator, Robert Naclerio, Professor, University of Chicago
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-224-A
Record Dates: First submitted 2010-10-28; First posted 2010-11-01 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allstate Nasal Spray (Active Comparator)
  Interventions: Device: Allstate Nasal Spray
- Placebo Nasal Spray (Placebo Comparator)
  Interventions: Device: Placebo Nasal Spray

INTERVENTIONS:
Device: Allstate Nasal Spray — Allstate Nasal Spray, two sprays (total 100 microliters) in each nostril.
  Arms: Allstate Nasal Spray
Device: Placebo Nasal Spray — 2 sprays in each nostril
  Arms: Placebo Nasal Spray

SUMMARY:
The purpose of this study is to see whether Allstate Nasal Spray when given in the nose is safe and can reduce the signs and symptoms of allergic rhinitis (hayfever).

ELIGIBILITY:
Inclusion Criteria

1. Males and females between 18 and 55 years of age.
2. History of grass and/or ragweed allergic rhinitis for at least 2 years.
3. Positive skin test to grass and/or ragweed antigen within prior 12 months.
4. Positive response to screening nasal challenge.

Exclusion Criteria

1. Respiratory disease other than allergic rhinitis, allergic conjunctivitis and mild asthma.
2. Use of nasal steroids, antihistamines in the last 2 weeks.
3. Upper respiratory infection, sinusitis less than 2 weeks before screening.
4. Structural nasal abnormalities or nasal polyps on examination, nasal ulcer, frequent nose bleeding, recent nasal surgery or nasal trauma (within 90 days).
5. Having poorly tolerated previous administration of allergens
6. Nasolacrimal drainage system malfunctions.
7. Participation in other investigational therapy in the last 30 days.
8. Any systemic disorder or medication interfering with the study.
9. FEV1<80% of predicted at screening for subjects with mild asthma.
10. Presence of allergic rhinitis symptoms in the screening period with TNSS >3 at baseline)
11. Undergoing allergen desensitization therapy.
12. Current smokers or recent ex-smokers.
13. Not willing to give informed consent
14. Inability to understand the nature and requirements of the study, or to comply with the study procedures.
15. Any social or medical condition that, in the opinion of the investigator, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Number of sneezes and total nasal symptom score (TNSS) (sum of nasal stuffiness, nasal discharge, and nasal itching) (scale 0-3 for each symptom; total score 0-9) are co-primary endpoints. | 10 minutes following each nasal challenge

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Naclerio, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States